CLINICAL TRIAL: NCT03363542
Title: The Effects of Increased Fruits and Vegetables and/or Whole Grain Food Consumption on Cardio Metabolic Risk Factors of Subjects With Visceral Obesity
Brief Title: The Effects of Increased Fiber Diet Consumption on Outcomes of Subjects With Visceral Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: United Arab Emirates University (Other)
Responsible Party: Principal Investigator, Salah Gariballa, Professor, United Arab Emirates University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AJF201608
Record Dates: First submitted 2017-10-15; First posted 2017-12-06 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Visceral Obesity
MeSH Terms: conditions — Obesity, Abdominal | interventions — Fruit

STUDY DESIGN:
Intervention Model Description: diet rich in fruits, vegetables and/or whole-grain fiber
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fruits and vegetables rich diet (Active Comparator): dietary education to increase fruits and vegetable consumption
  Interventions: Dietary Supplement: fruits, vegetables and/or whole grain high fiber rich diet
- Whole grain fiber rich diet (Active Comparator): dietary education to increase whole grain fiber consumption
  Interventions: Dietary Supplement: fruits, vegetables and/or whole grain high fiber rich diet
- Fruits and vegetables and whole grain fiber rich diet (Active Comparator): dietary education to increase fruits and vegetable and whole grain fiber consumption
  Interventions: Dietary Supplement: fruits, vegetables and/or whole grain high fiber rich diet
- Control group (No Intervention): Routine care

INTERVENTIONS:
Dietary Supplement: fruits, vegetables and/or whole grain high fiber rich diet — Dietary education to Increase fruits, vegetables and/or high fiber intake
  Arms: Fruits and vegetables and whole grain fiber rich diet; Fruits and vegetables rich diet; Whole grain fiber rich diet

SUMMARY:
The investigators propose to undertake a controlled dietary intervention study in UAE subjects with visceral obesity to examine the feasibility of a diet rich in fruits, vegetables and/or whole-grain fiber in the UAE population. The research will also investigate the longer-term influence of increased fruits, vegetables and fiber consumption on health and its capacity to sustain lifestyle change.

DETAILED DESCRIPTION:
The United Arab Emirates (UAE) has one of the highest prevalence of obesity related diabetes mellitus in the World [3]. Visceral (abdominal) obesity is particularly common and more closely related to morbidity in the UAE. The investigators propose to undertake a controlled dietary intervention study in UAE subjects with visceral obesity, the aims of which are: (i) To examine the feasibility of a diet rich in fruits, vegetables and/or whole-grain fiber in the UAE population (ii) To examine the effects of increased fruits, vegetables and/or whole-grain fiber consumption on cardio metabolic risk factors (iii) To investigate the longer-term influence of increased fruits, vegetables and fiber consumption on health and its capacity to sustain lifestyle change. The proposed study will provide the scientific rationale and the methodology for improving the diet and promote healthy eating in the UAE population.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with visceral obesity (WC=>88 cm for women and =>92 cm for men).

Exclusion Criteria:

* Individuals with severe chronic clinical or psychiatric disease, 2) Participating in other intervention trials, have a special diet or taking supplements. Consent All volunteers will be required to provide informed written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Waist circumference in cm | baseline and 6 months
  Change in waist circumference

CONTACTS AND LOCATIONS:
Overall Officials: Salah Gariballa, MD, Principal Investigator — United Arab Emirates University
Locations (1):
- United Arab Emirates University, Al Ain City, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No